CLINICAL TRIAL: NCT02093130
Title: Twelve-Month, Double-blind, Placebo-Controlled Study of Pomegranate Juice in Normal Aging
Brief Title: Study of Pomegranate Juice on Memory in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Principal Investigator, Gary Small, MD, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-001644
Record Dates: First submitted 2014-03-14; First posted 2014-03-20 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Impact of Pomegranate Juice on Memory in Older Adults
Keywords: Double-blind Trial; Placebo-controlled; Pomegranate; Memory; Memory Impairment; Cognition; Ages 50-75
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate Juice (Experimental): Eight ounces of 100% Pomegranate Juice daily
  Interventions: Dietary Supplement: Pomegranate Juice
- Placebo (Placebo Comparator): Eight ounces of Placebo juice daily. The Placebo is engineered to look and taste the same as the Pomegranate Juice and contains the same vitamins and minerals as the Pomegranate Juice. Because the Placebo juice does not come from actual pomegranates, it does not contain the polyphenols contained in the Pomegranate Juice.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice
  Arms: Pomegranate Juice
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This project is designed to study whether pomegranate juice benefits cognitive abilities in middle-aged and older non-demented volunteers. Subjects will be randomly assigned to one of two treatment groups: either a placebo or the pomegranate juice. Subjects will drink eight ounces of the pomegranate juice or placebo daily for twelve months.

The investigators expect the people receiving the pomegranate juice to show better cognitive performance compared with those receiving a placebo after one, six, and twelve months. The investigators believe cognitive decline and treatment response will vary according to a genetic risk for Alzheimer's.

The investigators will study 212 non-demented subjects aged 50-75 years. Initially, subjects will undergo a clinical assessment, an MRI and a blood draw to determine genetic risk and to rule out other neurodegenerative disorders linked to memory complaints.

Subsequently, subjects will undergo the first memory (or neuropsychological) assessments. Following the first assessment, subjects will begin drinking the juice (either the pomegranate juice or the placebo). Subjects will undergo a brief memory test at one-month mark. At six months, subjects will have a second, full neuropsychological assessment. The final assessment will take place at the end of the study, the 12-month mark. Additional blood will be drawn at baseline and at 12 months and frozen to assess inflammatory markers if outcomes are positive.

In total, subjects will be expected to come to the University of California, Los Angeles (UCLA) for 5 visits during the course of 12-13 months.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the 12-month double-blind, placebo-controlled clinical trial of pomegranate extract.
* Nondemented subjects either those with normal cognition or with Mild Cognitive Impairment will be included.
* Age 50 to 75 years.
* No significant cerebrovascular disease: modified Ischemic Score of < 4
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Screening laboratory tests and EKG without significant abnormalities that might interfere with the study. If screening laboratory tests or EKG show abnormalities, subject must obtain written clearance from primary care physician before continuing in the study.

Exclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) or any other dementia (e.g., vascular, Lewy body, frontotemporal) (McKhann et al, 1984). Evidence of other neurological or physical illness that can produce cognitive deterioration. Volunteers with a history of stroke, Transient Ischemic Attack (TIA), carotid bruits, or lacunes on MRI scans will be excluded. Determination of dementia will be based on the clinical evaluation including assessment of functional abilities, and cognitive screening.
* Contraindication to the MRI including claustrophobia, metal in body, surgery within 60 days, certain implants or previous abnormal MRI results.
* Evidence of Parkinson's disease as determined by the motor examination (items 18-31) of the Unified Parkinson's Disease Rating Scale (Fahn et al, 1987).
* History of myocardial infarction within the previous year, or unstable cardiac disease.
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100).
* History of significant liver disease, clinically-significant pulmonary disease, or diabetes.
* Current diagnosis of any major psychiatric disorder.
* Current diagnosis or history of alcoholism or substance addiction.
* Regular use of any medication that may affect cognitive functioning including: centrally active beta-blockers, narcotics, Clonidine, anti-Parkinsonian medications, antipsychotics, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, or Warfarin.
* Occasional use of anxiety or sleeping medications known to cause cognitive dulling will be allowed, but discouraged: chloral hydrate, non-benzodiazepine hypnotics such as: Ambien (Zolpidem) and Lunesta; or benzodiazepines such as Ativan (Lorazepam), Xanax (Alprazolam), Klonopin (Clonazepam), and Restoril (Temazepam).
* Use of any of the following medications: Amitriptyline, Amiodarone, Desipramine, Fenofibrate, Flecainide, Fluconazole, Fluoxetine, Fluvastatin, Fluvoxamine, Isoniazid, Lovastatin, Ondansetron, Phenylbutazone, Probenecid, Sertraline, Sulfamethoxazole, Sulfaphenazole, Teniposide, Voriconazole, Warfarin, and Zafirlukast
* Use of cognitive enhancing supplements (e.g. Ginkgo biloba).
* Use of any supplement containing pomegranate or pomegranate juice.
* Use of any investigational drugs within the previous month or longer, depending on drug half-life.
* Pregnancy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in cognitive testing results from Baseline to 1, 6, and 12 months | 1 year
  Non-demented volunteers aged 50-75 who receive a daily dietary supplement of pomegranate juice will show improved cognitive performance compared to baseline versus those receiving a placebo after one, six, and twelve months.

SECONDARY OUTCOMES:
Correlation between cognitive change and genotype | 1 year
  Cognitive change in the pomegranate intervention group will vary according to genotypes found to influence age at dementia onset (e.g., apolipoprotein E [APOE] TOMM40).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Small, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Longevity Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Siddarth P, Thana-Udom K, Ojha R, Merrill D, Dzierzewski JM, Miller K, Small GW, Ercoli L. Sleep quality, neurocognitive performance, and memory self-appraisal in middle-aged and older adults with memory complaints. Int Psychogeriatr. 2021 Jul;33(7):703-713. doi: 10.1017/S1041610220003324. Epub 2020 Sep 28. PMID 32985406
- [Derived] Siddarth P, Li Z, Miller KJ, Ercoli LM, Merril DA, Henning SM, Heber D, Small GW. Randomized placebo-controlled study of the memory effects of pomegranate juice in middle-aged and older adults. Am J Clin Nutr. 2020 Jan 1;111(1):170-177. doi: 10.1093/ajcn/nqz241. PMID 31711104
- See also: UCLA Longevity Center — http://www.semel.ucla.edu/longevity